Aldeyra Therapeutics, Inc.

Statistical Analysis Plan
Protocol No: ADX-102-AC-017

Final: V1.0, 26Mar2021

# Statistical Analysis Plan

The INVIGORATE Trial: A Single-Center, Randomized, Double-Masked, Crossover Design, Vehicle-Controlled, Phase 3 Clinical Trial to Assess the Efficacy and Safety of Reproxalap Ophthalmic Solution (0.25%) Compared to Vehicle in Subjects with Seasonal Allergic Conjunctivitis Using the Environmental Exposure Chamber (EEC)

**Protocol Number:** ADX-102-AC-017

**Protocol Version and Date:** Version 6.0, 24Mar2021

**Sponsor:** Aldeyra Therapeutics, Inc

**Indication:** Allergic Conjunctivitis

Analysis Plan Date: 26Mar2021

**Analysis Plan Version:** Version 1.0

#### **CONFIDENTIAL**

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Aldeyra Therapeutics, Inc. is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

# **SPONSOR SIGNATURE PAGE**

Protocol Title: The INVIGORATE Trial: a single-center, randomized, double-

masked, crossover design, vehicle-controlled, phase 3 clinical trial to assess the efficacy and safety of reproxalap ophthalmic solution (0.25%) compared to vehicle in subjects with seasonal allergic conjunctivitis using the environmental exposure chamber (EEC)

**Protocol Number:** ADX-102-AC-017

**Author:** 

**Sponsor:** Aldeyra Therapeutics, Inc.

131 Hartwell Avenue, Suite 320

Lexington, MA 02421

By signing this document, I acknowledge that I have read the document and approve of the planned statistical analyses described herein. I agree that the planned statistical analyses are appropriate for this study, are in accordance with the study objectives, and are consistent with the statistical methodology described in the protocol and all applicable regulatory guidance and guidelines.

| Approver: |
|-----------|

# **Table of Contents**

| SP | ONSO | R SIGNATURE PAGE | 2 |
|-----|-------|------------------------------------------------|----|
| LIS | ST OF | TABLES | 5 |
| AE | BREV | /IATIONS | 6 |
| 1. | INTR | RODUCTION | 7 |
| 2. | STUI | DY DESIGN | 7 |
| | 2.1 | OVERVIEW OF STUDY DESIGN | 7 |
| | 2.2 | Sample Size | 11 |
| | 2.3 | Randomization and Masking | 12 |
| | | 2.3.1 Randomization | 12 |
| | | 2.3.2 Masking | 12 |
| 3. | STUI | DY OBJECTIVES AND ENDPOINTS | 12 |
| | 3.1 | Primary Objective | |
| | 3.2 | Endpoints Assessment | 12 |
| | | 3.2.1 Clinical Trial Assessments and Endpoints | 12 |
| | | 3.2.2 Efficacy Endpoints | |
| 4. | DEFI | INITIONS AND CONVENTIONS FOR DATA HANDLING | |
| | 4.1 | Definition of Baseline | |
| | 4.2 | Handling of Missing Data | |
| | 4.3 | Unscheduled Visits for Safety Analysis | |
| | 4.4 | Handling of Partial Dates for Medications | |
| | 4.5 | Handling Partial Dates for Adverse Events | |
| 5. | ANA | LYSIS POPULATIONS | |
| | 5.1 | Enrolled Population | 14 |
| | 5.2 | Safety Population | |
| | 5.3 | Intent-to-Treat (ITT) Population | |
| | 5.4 | Completer Population | |
| | 5.5 | Per-Protocol (PP) Population | |
| | 5.6 | Application of Analysis Population | |
| 6. | | TISTICAL CONSIDERATIONS | |
| | 6.1 | General Statistical Procedures | |
| | 6.2 | Subject Disposition | |
| | 6.3 | Extent of Study Drug Exposure | |
| | 6.4 | Protocol Deviations | |
| | 6.5 | Demographic and Baseline Characteristics. | |
| | 6.6 | Medical and Social History | |
| | 6.7 | Prior and Concomitant Medications | |
| 7. | | y Analysis | |
| | 7.1 | Ophthalmic Examination Findings | |
| | 7.2 | Adverse Events | |
| | 7.3 | Clinical Laboratory Tests | 20 |

| Aldeyra Therapeutics, Inc. Protocol No: ADX-102-AC-017 | | Statistical Analysis Plan | |
|---|---|---|---|
| | | Final: V1.0, 26Mar2021 | |
| | 7.4 | Vital Signs | 21 |
| 8. | Efficacy Analysis | | 21 |
| | 8.1 | Primary Efficacy Analysis | 21 |
| | 8.2 | Key and Secondary Efficacy Analysis | 22 |
| 9. | Appe | endix | 24 |

Aldeyra Therapeutics, Inc.

Protocol No: ADX-102-AC-017

Statistical Analysis Plan
Final: V1.0, 26Mar2021

# LIST OF TABLES

| Table 1: Schedule of Events and Assessments | 8 |
|-----------------------------------------------|----|
| Table 2. Application of Populations on Tables | 15 |

# **ABBREVIATIONS**

| Abbreviation | Explanation |
|--------------|----------------------------------------------|
| AE | Adverse Event |
| AR1 | First-order Autoregressive |
| ATC | Anatomical Therapeutic Chemical |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CS | Compound Symmetric |
| EEC | Environmental Exposure Chamber |
| IOP | Intraocular Pressure |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model Repeated Measures |
| NCT | Non-Contact IOP Tonometry |
| PP | Per-Protocol |
| PT | Preferred Term |
| SD | Standard Deviation |
| SLE | Slit Lamp Examination |
| SOC | System Organ Class |
| TEAE | Treatment-Emergent Adverse Event |
| TOSS | Total Ocular Symptom Score |
| VA | Visual Acuity |
| WHO | World Health Organization |
| WOCBP | Women of Childbearing Potential |

#### 1. INTRODUCTION

This statistical analysis plan is designed to outline the statistical methods for protocol ADX-102-AC-017:

"The INVIGORATE Trial: A single-center, randomized, double-masked, crossover design, vehicle-controlled, Phase 3 clinical trial to assess the efficacy and safety of reproxalap ophthalmic solution (0.25%) compared to vehicle in subjects with seasonal allergic conjunctivitis using the environmental exposure chamber (EEC)"

This document has been prepared based on protocol amendment version 6.0 dated 24 March 2021

#### 2. STUDY DESIGN

#### 2.1 OVERVIEW OF STUDY DESIGN

The double-masked, vehicle-controlled, randomized, two-way crossover clinical trial allows for the testing of Reproxalap Ophthalmic Solution (0.25%) versus Vehicle Ophthalmic Solution in subjects with ragweed-induced allergic conjunctivitis in the Environmental Exposure Chamber (EEC).

The clinical trial consists of four visits to the clinic (one Medical Screening visit, one Screening EEC visit, and two EEC treatment visits). The EEC sessions will be separated by an approximate two-week washout period to ensure adequate elimination of responses caused by allergen exposure in the EEC and allow the recuperation of mast cells.

The EEC clinical research facility is a room designed with the capacity and control mechanisms to expose participants to airborne ragweed pollen grains and maintains target temperature and relative humidity throughout.



The controlled pollen challenge, over time, allows evaluation of subject responses at any time-point throughout the challenge process.

Aldeyra Therapeutics, Inc.

Statistical Analysis Plan
Protocol No: ADX-102-AC-017

Final: V1.0, 26Mar2021

Figure 1: Study Design



Eligible subjects will be randomized 1:1 to one of two treatment sequences of AB or BA where:

- Treatment A: Reproxalap Ophthalmic Solution (0.25%)
- Treatment B: Vehicle Ophthalmic Solution

Approximately 126 subjects (approximately 63 per treatment sequence) will be enrolled and will follow the schedule for assessments (Table 1).

**Table 1: Schedule of Events and Assessments** 



At the **Medical Screening Visit (Visit 1)**, subjects will undergo the informed consent process, and information about demographics, baseline characteristics, medical history, social history, physical examination will be performed and concomitant medication will be collected. Vital signs and samples for standard clinical safety laboratory tests will be obtained. A urine pregnancy test will be administered to women of childbearing potential (WOCBP).

Subjects will undergo ophthalmic examinations (Snellen VA, SLE, NCT, and a dilated fundus examination) to ensure initial eligibility criteria are met. A skin prick test for a panel of test allergens will be conducted; results must be positive (i.e., a wheal that is 3 mm greater than the negative control) for at least one test allergen and must include ragweed in order to proceed to Visit 2.

At all EEC sessions, assessments of ophthalmic evaluations will be collected

In the event of an failure, paper diary cards will be used as a back-up to collect symptom scores. For subject-reported symptoms of ocular itching, a standard 9 point (i.e., 0-4 with 0.5 unit increments) scale will be employed. For staff-assessed grading of conjunctival redness, a standard 9-point (i.e., 0-4 with 0.5 unit increments) will be employed.

| - | herapeutics, Inc.<br>No: ADX-102-AC-017 | Statistical Analysis Plan<br>Final: V1.0, 26Mar2021 |
|---|---|---|
| collect A | EC Screening Visit (Visit 2), qualified site staff will update concord AEs, as applicable and perform tests for vital signs. A urine pered to WOCBP. Fundus exam, Snellen VA, SLE, subject rating of conjunctival redness will be performed to ensure the anterior | regnancy test will be of symptoms, and staff |
| Visit 2 P | Pre-EEC entry (Baseline): | |
| 1) S | subject assessment for ocular itching and tearing will be recorded, and | |
| 2) S | taff-assessed conjunctival redness will be recorded. | |
| Visit 2 P | Post-EEC entry: | |
| 1) S | subject assessment for ocular itching and tearing will occur | |
| 2) S | taff-assessed conjunctival redness will be recorded . | |

At the Randomization/Treatment EEC Session One (Visit 3), qualified site staff will update concomitant medications, collect AEs, as applicable and collect vital signs. A urine pregnancy test will be administered to WOCBP. Ophthalmic evaluations will be conducted (Fundus exam, Snellen VA, NCT SLE, subject rating of symptoms, and staff grading of conjunctival redness).

Subjects will be randomized to receive a first dose of either Reproxalap Ophthalmic Solution (0.25%) (Treatment A) or Vehicle Ophthalmic Solution (Treatment B). Qualified site staff will instill one drop of the randomized treatment into each eye at approximately time zero prior to entry to the EEC after all the pre-EEC assessments are done.

# **Visit 3 Pre-EEC entry (Baseline):**

| Aldeyra | Therapeutics, Inc. | Statistical Analysis Plan |
|---|---|---|
| Protocol | No: ADX-102-AC-017 | Final: V1.0, 26Mar2021 |
| 1) | Subject assessment for ocular itching and tearing will be recorded | |
| | and | |
| 2) | Staff-assessed conjunctival redness will be recorded | |
| Visit 3 | Post-EEC entry: | |
| 1) | Subject assessment for ocular itching and tearing will occur | |
| 2) | Staff-assessed conjunctival redness will be recorded | |
| At app | roximately 90-minutes post-EEC entry (and after subject assessed ito | thing and tearing and |
| staff as | ssessed conjunctival redness for all time-noints post first dose have | heen completed) a |

staff assessed conjunctival redness for all time-points post first dose have been completed), a second dose (one drop in each eye) of the same randomized treatment will be administered in each eye by the qualified site staff.

# Visit 3 Post-EEC exit (starting at approximately t = 215 minutes):

- 1) Subject assessed ocular itching and tearing will continue .
- 2) Staff assessed conjunctival redness will continue to be recorded post-EEC exit .

Subjects will be asked to return in at least two weeks for Visit 4.

At the **Treatment EEC Session Two (Visit 4)**, all procedures performed at Visit 3 will be repeated except that each subject will be given a different treatment dependent on the treatment sequence the subject was randomized to [Reproxalap Ophthalmic Solution (0.25%) (Treatment A) or Vehicle Ophthalmic Solution (Treatment B)].

Before EEC entry, a urine pregnancy test will be administered to WOCBP.

Subjects will undergo ophthalmic examinations (Snellen VA, SLE, NCT, and a dilated fundus examination), clinical safety lab tests and vital signs will be collected to ensure safety prior to exit of the clinical trial.

#### 2.2 Sample Size

Approximately 670 subjects with ragweed-induced, moderate-to-severe allergic conjunctivitis will be screened in the EEC in order to randomize approximately 126 subjects, and for 100 subjects to

Statistical Analysis Plan Final: V1.0, 26Mar2021

complete the study. Approximately sixty-three (63) subjects will be assigned to each of two (2) treatment sequences, AB and BA.



#### 2.3 Randomization and Masking

#### 2.3.1 Randomization

Eligible subjects will be randomized 1:1 to one of two treatment sequences of AB or BA where:

- Treatment A: Reproxalap Ophthalmic Solution (0.25%)
- Treatment B: Vehicle Ophthalmic Solution

Approximately 126 subjects (approximately 63 per treatment sequence) will be enrolled.

Each subject screened for the clinical trial will be assigned a unique subject number that will be used to identify the subject throughout subject participation in the clinical trial. If a subject fails to be randomized, the reason should be documented in the source documents and case report form (CRF). The subject will be considered a screen failure.

## 2.3.2 Masking

Investigators, qualified site personnel, and subjects will be masked to the investigational product (IP) administered. The Sponsor will also be masked to the IP administered until database lock.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

#### 3.1 Primary Objective

• To evaluate the efficacy and safety of Reproxalp Ophthalmic Solution (0.25%) compared to Vehicle Ophthalmic Solution for the treatment of allergic conjunctivitis using the EEC clinical trial design

#### 3.2 Endpoints Assessment

#### 3.2.1 Clinical Trial Assessments and Endpoints

- Ocular itching rated by the subject using a 9-point, discrete, 0-4 scale with 0.5 increments
- Tearing rated by the subject using a 4-point discrete 0-3 scale
- Ocular redness in the nasal and temporal conjunctiva separately in both eyes, based on a descriptive and photographic scale from 0-4 with 0.5 steps

• Total Ocular Symptom Score (TOSS): composite score of ocular itching (0-4), ocular tearing (0-3) and ocular redness (0-4) with a maximum score of 11 units

## 3.2.2 Efficacy Endpoints

#### 3.2.2.1 Primary Efficacy Endpoint

• Change from baseline in ocular itching score on a 9-point scale (0-4) from 110-210 minutes

#### 3.2.2.2 Key Secondary Endpoint

• Change from baseline in conjunctival redness on a 9-point scale (0-4) during the chamber (approximately 12 to 212 minutes)

### 3.2.2.3 Secondary Endpoints

- Change from baseline in tearing on a 4-point scale (0-3) during the chamber (approximately 10 to 210 minutes)
- Change from baseline in TOSS on an 11-point composite score (sum of maximum score of itching, tearing and redness) during the chamber (approximately 10 to 212 minutes)
- Safety Endpoints
- Ophthalmic examinations
  - Snellen visual acuity (VA)
  - Slit lamp examination (SLE)
  - Non-contact intraocular pressure tonometry (NCT)
  - Dilated fundus examination at screening Visit 1 and at Visit 4
  - Undilated fundus examination at Visits 2 and 3
- Adverse events
- Vital signs
- Clinical laboratory tests

#### 4. DEFINITIONS AND CONVENTIONS FOR DATA HANDLING

#### 4.1 Definition of Baseline

For Safety evaluations, baseline is defined as the last non-missing value measured prior to initiation of study drug.

### 4.2 Handling of Missing Data

Generally, imputation of missing data will not be performed.

# 4.3 Unscheduled Visits for Safety Analysis

All unscheduled visit values will be excluded from summary tables but will be included on data listing.

### 4.4 Handling of Partial Dates for Medications

When determining prior or concomitant medications, partial start dates of prior and concomitant medications will be assumed to be the earliest possible date consistent with the partial date.

For the purposes of analysis, incomplete medication start dates and stop dates will be imputed.

- If a medication start date is incomplete, January will be imputed for missing month and/or the first day of the month will be imputed for missing day.
- If a medication stop date is incomplete, December will be imputed for missing month and the last day of the month will be imputed for missing day.
- If the imputed medication stop date is after the date of study completion, the date of study completion will be used instead.

### 4.5 Handling Partial Dates for Adverse Events

When determining the treatment emergent AE, partial dates will be handled as follows.

- If the day of the month is missing, the onset day will be set to the first day of the month unless it is the same month and year as first dose date. In this case, the onset date will be assumed to be the first date of treatment.
- If the onset day and month are both missing, the day and month will be assumed to be January 1, unless the event occurred in the same year as the study treatment. In this case, the event onset will be coded to the day of treatment to conservatively report the event as treatment-emergent.
- A missing onset date will be coded as the day of treatment. If the resulting onset date is after a reported date of resolution, the onset date will be set equal to the date of resolution.
- Imputation of partial dates is used only to determine whether an event is treatmentemergent; data listings will present the partial date as recorded in the eCRF.

#### 5. ANALYSIS POPULATIONS

## 5.1 Enrolled Population

Enrolled Population includes all subjects with a signed informed consent form.

Aldeyra Therapeutics, Inc.

Statistical Analysis Plan
Protocol No: ADX-102-AC-017

Final: V1.0, 26Mar2021

### 5.2 Safety Population

Safety Population includes all randomized subjects who use at least one dose of investigational drug (Reproxalap Ophthalmic Solution or Vehicle Ophthalmic Solution), regardless of whether clinical trial assessments were performed.

# 5.3 Intent-to-Treat (ITT) Population

ITT Population includes all randomized subjects who use at least one dose of investigational drug and have any post-dose assessments. Subjects are evaluated according to the investigational drug treatment of the visit as per the randomized treatment sequence.

#### **5.4** Completer Population

Completer population will include all randomized subjects who received investigational drug dosing at all two EEC treatment visits.

### 5.5 Per-Protocol (PP) Population

Per-Protocol Population includes all subjects in Completer Population without a major deviation from the protocol.

## 5.6 Application of Analysis Population

Unless otherwise noted, the analysis populations that will be used for creating the summary tables of each type is provided in Table 2.



#### 6. STATISTICAL CONSIDERATIONS

All analyses described in this plan are considered a priori analyses in that they have been defined prior to locking the database. All other analyses, if any, designed subsequently to locking the database, will be considered post hoc analyses and will be described as exploratory analyses in the Clinical Study Report.

All summaries and statistical analysis will be performed

#### **6.1** General Statistical Procedures

Frequency distributions for categorical variables will be provided as number of patients in the category and the percentages of the total number of patients in the given population as noted. Percentages will be reported to one decimal place.

The descriptive statistics for continuous variables will be number of subjects (n), mean, standard deviation (SD), median, minimum and maximum. Mean and median will be reported to 1 more decimal place than the raw data, while the SD will be reported to 2 more decimal places than the raw data. Minimum and maximum will be reported the same as the original data.

All statistical tests will be two-sided with a significance level of 0.05 ( $\alpha = 0.05$ ) unless otherwise specified. Confidence interval (CI) for differences between treatment will be two-sided at 95% confidence interval.

P-value will be rounded to at most 3 decimal places and will be reported as < 0.001 if it is smaller than 0.001.

Unless otherwise specified, subjects' characteristics at baseline will be summarized by treatment sequences (Reproxalap 0.25%/Vehicle, Vehicle/Reproxalap 0.25%). Safety and efficacy will be summarized by treatment (Reproxalap 0.25%, Vehicle) where appropriate.

In general, all listings will be ordered by subject number and visit for available data unless otherwise specified in the text.

#### **6.2** Subject Disposition

Frequency and percentage of subject disposition will be summarized by treatment sequence and all subjects for Enrolled Population including:

- Number of subjects with screen failure
- Number of subjects randomized
- Number of subjects in each analysis population
- Number of subjects who completed each treatment
  - Reproxalap Ophthalmic Solution 0.25%
  - Vehicle Ophthalmic Solution
- Number of subjects only completed first treatment session

Percentage will be based on number of subjects randomized.

Study discontinuation will be summarized by treatment for Safety Population including:

- Number of subjects discontinued from study
- Reasons for study discontinuation

Aldeyra Therapeutics, Inc.

Statistical Analysis Plan
Protocol No: ADX-102-AC-017

Final: V1.0, 26Mar2021

- Subject request/withdrawal
- Adverse event
- Pregnancy
- Protocol violations
- Administrative reasons
- Sponsor termination
- Any sound medical reason
- Other

Percentage is based on number of subjects in Safety Population.

Subjects' disposition will be listed for Enrolled Population. In addition, subjects excluded from study will be listed for Enrolled Population.

## 6.3 Extent of Study Drug Exposure

Exposure of study drug will be listed for Safety Population.

#### 6.4 Protocol Deviations

Protocol deviations will be reviewed, assessed and documented by sponsor personnel before database lock.

Number and percentage of subjects with protocol deviation will be tabulated by treatment for Safety Population. The protocol deviations will be grouped into different categories which may include, but are not limited to:

- Missed visit
- Inclusion/Exclusion criteria
- Missed procedures/assessments
- Informed consent
- Documentation
- Study drug administration
- Safety
- Lack of compliance

All protocol deviations will be listed for Enrolled Population.

#### 6.5 Demographic and Baseline Characteristics

Subjects' demographic and baseline characteristics will be summarized by treatment sequence and for all subjects including:

- Age at screening (years). If not reported, calculated as integer of (date of informed consent signed date of birth)/365.25 and rounded to integer.
- Sex
- Race
- Ethnicity
- Height (cm)
- Weight (kg)
- BMI (body mass index, kg/m<sup>2</sup>), calculated as weight (kg) / height (m)<sup>2</sup>

Demographics and baseline characteristics will be listed for ITT Population.

## 6.6 Medical and Social History

Medical and social history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA)

The frequency count and percentage of patients experiencing any medical conditions will be tabulated by system organ classifications (SOC) and preferred term (PT) for each treatment. If a preferred term or system organ class was reported more than once for a subject, the subject would only be counted once in the incidence for that preferred term or system organ class.

Medical history data will be listed for ITT Population.

#### 6.7 Prior and Concomitant Medications

All medications will be coded according to the WHO drug dictionary which includes the WHO Drug Preferred Name and the ATC Classification Level 2 and 4.

Prior medications are medications used 30 days prior to consent to treat any medical conditions and will be documented at medical screening visit.

Concomitant medications are medications being taken on or after first dose the study drug. Medications taken 30 days prior to informed consent date and were ongoing on the date of the first dose will be considered concomitant medications. Medications with missing end date are assumed to be concomitant medications.

Prior and concomitant medications will be listed ONLY for ITT Population.

# 7. Safety Analysis

#### 7.1 Ophthalmic Examination Findings

Ophthalmic examination results will be summarized by anatomical location (eye) and side (left, right and both) at pre and post-EEC entry treatment sessions for Safety Population for following tests:

- Visual acuity measured using a Snellen eye chart
- Slit lamp examination (SLE)
- Non-contact intraocular pressure tonometry (NCT), measured using non-contact tonometry
- Fundoscopy including:
  - Dilated fundus examination at Visit 4
  - Undilated fundus examination at Visits 3

#### 7.2 Adverse Events

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary preferred term (PT) and system organ classification (SOC).

An AE will be considered treatment emergent (TEAE) if it begins or worsens in severity after the first dose of the study drug through 30 days after the last dose of study drug, or the date of initiation of another investigational agent or surgical intervention.

Drug-related TEAEs are defined as definitely related, possibly related, or probably related to study drug. Any AEs with missing relationship to study drug will be considered as related to study drug.

All TEAEs with start dates prior to first dose date in Visit 4 EEC Treatment Session will be classified as AEs occurred in Visit 3 EEC Treatment Session.

An overall summary for number of subjects with events in each treatment will be provided including:

- Number of subjects with at least one TEAE
- Number of subjects with at least one Ocular TEAE
- Number of subjects with at least one drug-related TEAE
- Number of subjects with at least one drug-related Ocular TEAE
- Number of subjects with at least one serious TEAE
- Number of subjects with at least one serious Ocular TEAE
- Number of subjects with at least one TEAE leading to study discontinuation
- Number of subjects with at least one Ocular TEAE leading to study discontinuation

An AE is classified as an ocular AE if system organ class is coded as eye disorders.

The following types of summary for each treatment will be provided. Summaries will be sorted by decreasing frequency of PT within SOC which will be sorted alphabetically.

- TEAEs by SOC and PT
- Ocular TEAEs by SOC and PT
- Non-Ocular TEAEs by SOC and PT
- TEAEs by Casualty, SOC and PT

- Ocular TEAEs by Casualty, SOC and PT
- Non-Ocular TEAEs by Casualty, SOC and PT
- Serious TEAE by SOC and PT
- Ocular Serious TEAE by SOC and PT
- Non-Ocular Serious TEAE by SOC and PT
- TEAE by SOC, PT and maximum Severity
- Ocular TEAE by SOC, PT and maximum Severity
- Non-Ocular TEAE by SOC, PT and maximum Severity
- TEAEs leading to study discontinuation by SOC and PT
- Ocular TEAEs leading to study discontinuation by SOC and PT
- Non-Ocular TEAEs leading to study discontinuation by SOC and PT

If a preferred term or system organ class was reported more than once for a subject, the subject would only be counted once in the incidence for that preferred term or system organ class.

- In the tabulation of TEAE by severity, only the most severe PT or SOC for each subject will be included. Missing severity will be counted as Severe.
- In the summary of drug-related TEAEs, the strongest relationship will in included.

Listing will be provided including for Safety Population:

- All AEs
- Serious TEAEs
- TEAEs leading to study discontinuation

# 7.3 Clinical Laboratory Tests

Standard clinical safety laboratory (chemistry and hematology) collected at the Medical Screening Visit (Visit 1) and the second Treatment EEC Session (Visit 4) as part of study exit procedures include following parameters:

- Hematology profile: hemoglobin, hematocrit, red blood cell (RBC) count, white blood cell (WBC) count, and absolute platelet count
- Serum chemistry profile: albumin, alkaline phosphatase (ALP), ALT (SGPT), AST (SGOT), BUN, calcium, carbon dioxide (CO2), chloride, total cholesterol, creatinine, creatinine phosphokinase (CPK), glucose, phosphate, potassium, sodium, total protein, and uric acid.

All laboratory tests including pregnancy testing will be provided. Separate listing will also be provided for clinically significant abnormal laboratory values.

## 7.4 Vital Signs

Vital sign assessments will be taken with the subject in the sitting or supine position after 5 minutes at rest and will include body temperature, pulse rate, blood pressure (BP), and respiratory rate (RR) prior to EEC entry and at end of Visit 4 prior to study exit.

Observed and changes from baseline for vital signs will be summarized by visit. Baseline is defined as the last non-missing measurement taken prior to the first dose.

Listing will be provided for ITT Population.

# 8. Efficacy Analysis

The efficacy evaluation will be performed to assess the activity of Reproxalap Ophthalmic Solution based on the subjects reported ocular itching using a standard 9-point scale (0-4 scale with 0.5-unit increments) and tearing on a standard 4-point (0-3 scale) and trained staff assessed conjunctival redness using a standard 9-point scale (0-4 scale with 0.5 unit increments).

For all staff assessed and subject reported symptoms where values from both eyes are obtained at the same timepoint, the average score from both eyes will be used for analysis.

The following analysis will be performed for all efficacy endpoints using ITT Population:

- Observed and changes from baseline by visit and treatment
- Analysis using Mixed Model Repeated Measures (MMRM) using all available data collected during the EEC
- Plots for mean score over time, and mean changes of score from baseline over time

The onset of action time point and the duration of action will be reported for each efficacy endpoint whenever applicable. Duration of action will be the longest (in minutes) series of time points over which majority is statistically significant in favor of test drug, including the first and last time points in the series. Onset of action will be the first time point in the duration series. If two or more duration series are equivalent in length (in minutes), then the onset will be the first time point in the series that occurs earliest.

Subjects' assessment at Screening EEC and Post-EEC exit time points will be listed ONLY. All efficacy data will be listed for ITT Population.

## 8.1 Primary Efficacy Analysis

The primary efficacy endpoint is the change from baseline (pre-dose) in ocular itching scores on a 9-point scale (0-4 scale with 0.5-unit increments) from 110-212 minutes between Reproxalap Ophthalmic Solution (0.25%) and vehicle.

Observed and changes from baseline duration treatment period will be summarized by visit and treatment for ITT, PP, and Completer populations.

Primary efficacy analyses will be carried out in the ITT population. Supportive analyses for primary efficacy endpoint will also be provided using the PP population and the Completer population if more than 10% of ITT population is excluded from PP population.

The treatment comparison will be performed by using a Mixed Model Repeated Measures (MMRM) approach for a crossover study with 2 treatment periods (Visit 3 treatment EEC Session One and Visit 4 treatment EEC Session Two)



Reproxalap Ophthalmic Solution will be claimed to be better than Vehicle if the estimated change of ocular itch score from baseline based on MMRM model in the Reproxalap group is statistically lower than that of the Vehicle group

If the MMRM model does not converge with any correlation structure, then a within-subject t-test (baseline-adjusted, if useful) will be used to compare the score difference across treatment groups at each time point.

## 8.2 Key and Secondary Efficacy Analysis

The key secondary efficacy endpoint is

• Change from baseline in conjunctival redness on a 9-point scale (0-4) during the chamber (approximately 10 to 210 minutes)

The secondary efficacy endpoints are

Statistical Analysis Plan Final: V1.0, 26Mar2021

Aldeyra Therapeutics, Inc. Protocol No: ADX-102-AC-017

- Change from baseline in tearing on a 4-point scale (0-3) during the chamber (approximately 10 to 210 minutes)
- Change from baseline in TOSS on an 11-point composite score (sum of itching, tearing, and redness) during the chamber (approximately 10 to 210 minutes)

TOSS will be derived as the sum of ocular itching, conjunctival redness and tearing symptoms at each time point.

Observed and changes from baseline duration treatment EEC session will be summarized by visit and treatment for ITT population.

All secondary efficacy endpoints will be analyzed using a similar approach as the primary efficacy variable for the ITT Population. Reproxalap Ophthalmic Solution will be claimed to be better than Vehicle on secondary efficacy endpoints if the estimated overall corresponding changes from baseline score from MMRM model in the Reproxalap group is statistically lower than that of the Vehicle group during the chamber (approximately 10 to 210 minutes).

Statistical Analysis Plan Final: V1.0, 26Mar2021

